CLINICAL TRIAL: NCT02764476
Title: Safety and Feasibility of Virtual Reality Therapy for Functional Neurological Symptom/Conversion Disorder
Brief Title: Embodied Virtual Reality Therapy for Functional Neurological Symptom/ Conversion Disorder
Acronym: VR4FND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID emergency
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kim Bullock, MD, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36842
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Conversion Disorder; Psychogenic Movement Disorder; Functional Movement Disorder; Functional Neurological Disorder; Non-epileptic Seizures
Keywords: psychogenic; non-epileptic seizures; functional neurological symptom disorder; PNES; PMD; virtual reality; 3D augmented reality; mirror therapy
MeSH Terms: conditions — Conversion Disorder; Seizures

STUDY DESIGN:
Intervention Model Description: Single blinded randomized control trial for 8 weeks, then control group will be offered active treatment if desired.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality Therapy (Experimental): Eight 30 minute sessions of embodied virtual reality therapy with use of a body transfer experience into an egocentric perspective avatar that encourages motor activity and desensitization to emotional cues.
  Interventions: Other: Embodied Virtual Reality Therapy
- Control (Active Comparator): Eight 30 minute sessions of virtual reality therapy.
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Embodied Virtual Reality Therapy — Participants will be asked to play a game in Stanford's Virtual Reality Human Interaction Lab that engages visual pathways and involves body tracking and controlled sensory feedback reinforcing movement in real and virtual time by immersive head mounted displays. This game will have subjects fully embody and inhabit an avatar from an egocentric perspective. In addition, over consecutive sessions subjects will be asked to use a mobile smart phone based virtual reality program designed to deliver various and customized emotionally provocative stimuli.
  Arms: Virtual Reality Therapy
Other: Virtual reality — Participants will be asked to play a game in Stanford's Virtual Reality Human Interaction Lab that engages visual pathways.
  Arms: Control

SUMMARY:
The purpose of this study is to design and test the safety and feasibility of virtual reality technologies and experiences of egocentric avatar embodiment in the application of physical and cognitive behavior therapy in functional neurological symptom/conversion disorder. Investigators hypothesize that patients will safely use and accept this modality of treatment and will show evidence of a decrease in symptom frequency.

DETAILED DESCRIPTION:
This is a treatment development trial, participants randomly assigned to active treatment will be enrolled in embodied Virtual Reality therapy. The therapy will be based on principals of exposure and behavioral shaping therapies and mirror visual feedback therapy. The therapy will be delivered over 8 sessions and modified as indicated by clinical feedback. A fixed protocol will be developed with exact methods to be used to be determined. After a fixed protocol has been established, a treatment manual will be created to use in further controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years, who are diagnosed with functional neurologic symptom or conversion disorder. If diagnosis of seizure type then video EEG with diagnosis confirmed by board-certified neurologist with subspecialty training in epilepsy and clinical neurophysiology using the criteria of the International Classification of the Epilepsies is required. If diagnosis of motor type, documented and clinically established levels of diagnostic certainty (Williams,1995) confirmed by 2 neurologists is required.
* Participants must have at least one symptom per month in the month prior to enrollment
* Fluency in English spoken language

Exclusion Criteria:

* Nonfluency or inability to communicate in English spoken language
* Inability to participate or attend biweekly 30 minute session over 14 weeks
* Frank psychosis
* Active self harm urges
* Serious medical illness
* Active substance or alcohol use or dependence that could interfere with participation
* Diagnoses of mental retardation, dementia or delirium
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Adherence | Number of sessions attended over 12 weeks
  Number of sessions attended over 12 weeks recorded by therapist

SECONDARY OUTCOMES:
General Self-Efficacy Scale | baseline, biweekly for 6weeks, then 6,9,12 months
  self-report
Global Assessment of Functioning (GAF) | baseline, 6weeks, then 6,9,12 months
  physician administered Global Assessment of Functioning (GAF) is a numeric scale (1 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults
Generalized Anxiety Disorder 7-item (GAD-7) scale | baseline, biweekly for 6weeks then 6,9,12 months
  A 7 item self-complete questionnaire with very good sensitivity (89%) and specificity (82%) for Generalised Anxiety Disorder (GAD)
Patient Health Questionnaire-9 (PHQ-9) | baseline, biweekly for 6weeks then 6,9,12 months
  self-report
Oxford Handicap Scale | baseline, 6weeks, then 6,9,12 months
  physician administered
Frequency and severity of functional symptoms | baseline, biweekly for 6 weeks then 6,9,12 months
  self-report weekly log format
Frequency of adverse events | baseline, biweekly for 6 weeks then 6,9,12 months
  physician and subject report

CONTACTS AND LOCATIONS:
Overall Officials: Kim D Bullock, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bullock K, Won AS, Bailenson J, Friedman R. Virtual Reality-Delivered Mirror Visual Feedback and Exposure Therapy for FND: A Midpoint Report of a Randomized Controlled Feasibility Study. J Neuropsychiatry Clin Neurosci. 2020 Winter;32(1):90-94. doi: 10.1176/appi.neuropsych.19030071. Epub 2019 Nov 5. PMID 31687867
- See also: Midway point results — https://pubmed.ncbi.nlm.nih.gov/31687867/